CLINICAL TRIAL: NCT05775224
Title: ASH Research Collaborative Data Hub Protocol: A Multi-Center Data Hub of Individuals Living With Hematologic Disease
Brief Title: ASH Research Collaborative Data Hub
Status: Enrolling by invitation | Type: Observational
Sponsor: ASH Research Collaborative (Other)
Responsible Party: Sponsor
Other Study IDs: 20181051
Record Dates: First submitted 2023-01-13; First posted 2023-03-20 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Multiple Myeloma
Keywords: SCD; Sickle Cell; Myeloma
MeSH Terms: conditions — Anemia, Sickle Cell; Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sickle Cell Disease
- Multiple Myeloma

SUMMARY:
Benign and malignant hematologic diseases are relatively rare conditions within the spectrum of medical practice in any one site of care. Nonetheless, recent research in hematologic conditions from basic, translational, clinical and population perspectives offer the possibility of improving the way that these diseases are treated, and the outcomes experienced by patients. A repository that aggregates and validates this data across institutions and other practice settings is needed in order to identify variation in care, new findings, and further research.

DETAILED DESCRIPTION:
The ASH Research Collaborative (ASH RC) is a non-profit organization established by the American Society of Hematology (ASH) in 2018 that aims to improve the lives of those affected by blood diseases by fostering collaborative partnerships to accelerate progress in hematology. The foundation of the ASH RC is its Data Hub, a technology platform that facilitates the exchange of information by aggregating in one place, and making available for inquiry, research-grade data on hematologic diseases. In 2019, ASH RC launched its first research initiative, the Sickle Cell Disease (SCD) Clinical Trials Network (CTN), with the goal of optimizing SCD clinical research operations. As part of its core functions, the SCD-CTN leverages the Data Hub to collect key information and identify gaps that will help advance SCD research and treatment.

The primary goal of the Data Hub is to further the scientific knowledge base for the diagnosis, understanding, and management of benign and malignant hematologic conditions by assembling data collected in routine clinical care and closed clinical trials. Secondary goals are to characterize and study practice patterns for benign and malignant hematologic conditions in clinical practice, and to aggregate patient-reported data to further understand and improve the patient experience. These objectives will be fulfilled by amassing data from patients' electronic medical records and other data sources within institutions and networks to support prospective data collection efforts, such as those that include patient reported outcomes.

ELIGIBILITY:
To be included in the Data Hub, patients must have documented sickle cell disease and/or active multiple myeloma since 2015.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There will be no discrimination or bias with respect to inclusion on the basis of sex, race, or religion.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2099-04-29 (Estimated); Study Completion 2099-04-29 (Estimated)

PRIMARY OUTCOMES:
Data Collection | 50 year recruitment period (there will be continuous subgroup analyses through study completion)
  Aims of the Data Hub include collecting clinical data to gain further insights about diagnosis, treatment, prognosis, and risk factors of hematologic disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- ASH Research Collaborative, Washington D.C., District of Columbia, United States